CLINICAL TRIAL: NCT07023042
Title: Treatment of Kinesio-taping Versus Usual Care for Patients of Malignant Bowel Obstruction and Ascites With Persistent Severe Symptoms After Surgery, Medication and Nasogastric Tube: a Randomized Controlled Trial
Brief Title: Kinesio-Taping vs. Usual Care for Malignant Bowel Obstruction With Ascites
Acronym: KTMBO-RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202502118RINB
Record Dates: First submitted 2025-06-08; First posted 2025-06-15 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Malignant Bowel Obstruction; Ascites; Advanced Cancer
Keywords: Kinesio taping; Palliative care; Adjuvant therapy; Non-pharmacological intervention; Malignant Bowel Obsruction; Advanced Cancer; dmonton Symptom Assessment System; Symptom management
MeSH Terms: conditions — Ascites

STUDY DESIGN:
Intervention Model Description: This is a parallel assignment, randomized controlled trial with two arms: an intervention group receiving abdominal Kinesio-taping in addition to standard care, and a control group receiving standard care only. Participants are randomly assigned (1:1) to one of the two groups. No crossover or sequential treatment is planned. All outcome measures are assessed at baseline and three days after intervention.
Masking Description: No masking is used in this study because the nature of the intervention (abdominal Kinesio-taping) does not allow for blinding of participants or care providers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio taping Group (Experimental): Participants receive standard care for malignant bowel obstruction and ascites, plus abdominal Kinesio-taping applied by trained professionals according to a standardized protocol.
  Interventions: Other: Abdominal Kinesio taping
- Control Group (Active Comparator): Participants receive standard care for malignant bowel obstruction and ascites without Kinesio taping.
  Interventions: Other: Standard Care Arm

INTERVENTIONS:
Other: Abdominal Kinesio taping — Application of medical-grade Kinesio tape (NKH-50R) to the abdomen using a standardized circular technique, in addition to standard care for malignant bowel obstruction and ascites. Tape is applied by trained professionals after a skin sensitivity test and changed every three days or as needed. The procedure avoids open wounds and tumor sites. Participants and caregivers are educated on tape care and removal.
  Other Names: Kinesio taping; KT; Kinesiotaping; Kinesiology taping; Kinesiology tape; K-active tape
  Arms: Kinesio taping Group
Other: Standard Care Arm — Standard palliative care for malignant bowel obstruction and ascites, including symptom management, nutritional support, and medical treatment according to institutional protocols.
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to find out whether abdominal Kinesio-taping is a feasible and effective way to relieve symptoms in patients with malignant bowel obstruction and ascites who still have severe symptoms after surgery, medication, or nasogastric tube treatment.

The main questions it aims to answer are:

* Can abdominal Kinesio-taping reduce the severity of symptoms, such as abdominal pain, bloating, and nausea, in these patients?
* Is abdominal Kinesio-taping a safe and practical treatment option for this patient group?

Participants in this study are adults with cancer who have been diagnosed with malignant bowel obstruction and ascites, and whose symptoms have not improved after standard medical treatments. People who are allergic to tape, have abdominal wounds, are pregnant, or are unable to provide consent will not be included.

Participants will be randomly assigned to one of two groups:

* The Kinesio-taping group will receive standard care for malignant bowel obstruction plus abdominal Kinesio-taping, applied by trained professionals using a standardized procedure.
* The control group will receive standard care only.

The main outcomes measured will be changes in symptom severity using the Edmonton Symptom Assessment System (ESAS) modified for ascites, as well as abdominal girth and pain medication use. Symptoms and side effects will be closely monitored to ensure safety.

The information from this study may help determine whether Kinesio-taping can be an additional, safe, and effective option for managing symptoms in patients with advanced cancer who have malignant bowel obstruction and ascites.

DETAILED DESCRIPTION:
Malignant bowel obstruction (MBO) with ascites is a common and severe complication among patients with advanced intra-abdominal or retroperitoneal malignancies. Standard management of MBO includes surgery, medical therapy (such as antiemetics, corticosteroids, or octreotide), and decompression using nasogastric tubes. However, many patients continue to experience distressing symptoms-such as persistent abdominal pain, nausea, vomiting, and bloating-despite aggressive treatment. These symptoms contribute to significant discomfort, reduced quality of life, and poor prognosis in patients with advanced cancer.

Kinesio-taping is an elastic, waterproof adhesive strip designed to mimic the properties of skin and soft tissue. It is widely used in rehabilitation and sports medicine for its potential to reduce pain, improve circulation, and provide mechanical support. The mechanism is thought to involve stimulation of cutaneous mechanoreceptors, improved lymphatic drainage, and modulation of muscle activity. While Kinesio-taping has shown benefits in managing lymphedema and musculoskeletal pain, its application in patients with MBO and ascites is not well-studied. Existing evidence is mostly limited to case reports and studies in other patient populations.

This randomized controlled trial aims to evaluate whether abdominal Kinesio-taping, in addition to standard care, can safely and effectively reduce symptom burden in adult cancer patients with MBO and ascites whose symptoms persist after conventional treatment. The trial is conducted at a single tertiary medical center. Eligible patients are randomized in a 1:1 ratio to either the intervention group (standard care plus Kinesio-taping) or the control group (standard care alone). The Kinesio-taping protocol uses an FDA-approved medical-grade tape (NKH-50R) and follows a standardized application technique. Prior to the first application, all patients in the intervention group undergo a skin sensitivity test. The tape is applied in a circular pattern around the umbilicus, with specific attention to avoiding tumor sites and open wounds, and removed using techniques designed to minimize skin trauma.

All participants continue to receive standard care for MBO, including pain management, fluid and electrolyte support, and palliative interventions as appropriate. Data are collected at baseline and three days after intervention. The primary outcome is change in symptom severity, measured by the Edmonton Symptom Assessment System modified for ascites (ESAS:AM). Secondary outcomes include changes in abdominal girth and dosage of analgesic medications. Safety is monitored through daily assessment for skin reactions or other adverse effects.

This study is designed with rigorous attention to ethical conduct and data privacy. All participant information is de-identified and securely stored, and only authorized research personnel have access. The anticipated sample size is 40 participants, with randomization stratified by baseline symptom severity to ensure balanced allocation. Data will be analyzed using appropriate statistical methods, including independent t-tests and generalized estimating equations for repeated measures.

If proven effective and safe, Kinesio-taping could offer a non-invasive, low-cost, and easily administered adjunct to standard palliative care for patients with malignant bowel obstruction and ascites, potentially empowering both patients and caregivers with a new option for symptom relief.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Histologically confirmed intra-abdominal or retroperitoneal malignancy.
* Diagnosis of malignant bowel obstruction with ascites located below the ligament of Treitz.
* Persistent severe symptoms (such as pain, bloating, nausea, vomiting) after surgery, medication, or nasogastric tube treatment.
* Able to communicate in Mandarin or Taiwanese.
* Capable of providing informed consent.

Exclusion Criteria:

* Presence of significant abdominal wounds that preclude application of Kinesio tape.
* Known allergy or hypersensitivity to Kinesio tape.
* Pregnancy.
* Lack of decision-making capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2026-06-06 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in symptom severity score using the Edmonton Symptom Assessment System-Ascites Modification (ESAS:AM) | Baseline and 3 days after intervention
  Symptom severity will be measured using the ESAS:AM, which includes 11 items evaluating abdominal pain, bloating, nausea, and other symptoms related to malignant bowel obstruction and ascites. Each item is scored on an 11-point numeric rating scale (0-10), and the average score will be used for analysis. The primary outcome is the change in average symptom severity score from baseline to Day 3 after intervention.

SECONDARY OUTCOMES:
Change in abdominal girth | Baseline and 3 days after intervention
  Abdominal circumference will be measured in centimeters at the level of the umbilicus using a standard measuring tape. The primary comparison is the change in abdominal girth from baseline to Day 3 after intervention.
Change in analgesic medication use | Baseline and 3 days after intervention
  The total dose of analgesic medications (including morphine, fentanyl, oxycodone, and corticosteroids) administered to each participant will be recorded. The outcome is the change in total analgesic dose from baseline to Day 3 after intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to protect patient privacy and comply with local regulations